CLINICAL TRIAL: NCT00734916
Title: Immune Modulation by Omega-3 Versus Omega-6 Based Parenteral Lipids in Healthy Volunteers
Brief Title: Immune Modulation by Parenteral Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: M.W.J. Versleijen, MD, MSc and G.J.A. Wanten, MD, MSc, PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GW/MV/20307; CMO 2008/140
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Infections; Total Parenteral Nutrition
Keywords: total parenteral nutrition; infections; Infectious complications related to parenteral nutrition
MeSH Terms: conditions — Infections; Hyperphagia | interventions — fish oil triglycerides; soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Omegaven 10%
  Interventions: Dietary Supplement: Parenteral lipid emulsion (Omegaven)
- 2 (Active Comparator): Intralipid 10%
  Interventions: Dietary Supplement: Parenteral lipid emulsion (Intralipid)
- 3 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Parental lipid emulsion (Saline 0.9%)

INTERVENTIONS:
Dietary Supplement: Parenteral lipid emulsion (Omegaven) — Omegaven 10%, 0.2g/kg/hr i.v.during 1 hour on 3 consecutive days
  Other Names: Omegaven 10%, Fresenius Kabi, Bad Homburg Germany
  Arms: 1
Dietary Supplement: Parenteral lipid emulsion (Intralipid) — Intralipid 10%, 0.2g/kg/hr i.v. during 1 hour on 3 consecutive days
  Other Names: Intralipid 10%, Fresenius Kabi, Bad Homburg Germany
  Arms: 2
Dietary Supplement: Parental lipid emulsion (Saline 0.9%) — Placebo (Saline 0.9%), same volume/hr as lipid emulsions
  Other Names: lipid free control
  Arms: 3

SUMMARY:
Immune modulating properties of parenteral lipid emulsions seem to contribute to the increased risk for infections which remains associated with the use of total parenteral nutrition. Emulsions based on soy bean oil (SO) are the oldest and still most widely used lipid source in TPN formulations but their high content of omega-6 polyunsaturated fatty acids (PUFAs) may be a drawback. Fish oil-based lipid emulsions (FO), rich in omega-3 PUFAs, has been approved for parenteral nutrition in many countries. Mainly retrospective studies on clinical outcomes in septic and postoperative patients have suggested clinical benefits with the inclusion of FO in parenteral nutrition regimens. The exact mechanisms behind the beneficial immunological effects of parenteral FO have, however, not yet been elucidated.

Objective:

To evaluate the effects of intravenous infusion of a FO-based lipid emulsion and a SO-based emulsion on immune function as evidenced by effects on peripheral blood leukocyte counts and functions and on the susceptibility to oxidative stress.

Study design:

Randomized placebo controlled cross-over pilot study with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yrs of age)
* Healthy
* Willingness to give written informed consent

Exclusion Criteria:

* Smoking > 5 cigarettes/day
* Diet with > 2 portions of fatty fish per day
* Use of oral fish oil or vitamin substrates
* History of metabolic disorder (especially diabetes or lipid disorders)
* History of allergic, inflammatory of immunological disease
* History of pulmonary, cardiovascular, renal or hematological disease
* Medication use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
leukocyte counts | T=0, T=4 days, T=11 days
leukocyte functions | T=0, T=4 days and T=11 days
(anti-)oxidant status | T=0, T=4 days, T=11 days

SECONDARY OUTCOMES:
plasma and leukocyte cell membrane (phospho)lipid composition. | T=0, t=4 and T=11 days

CONTACTS AND LOCATIONS:
Overall Officials: Geert JA Wanten, MD, MSc, PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands